CLINICAL TRIAL: NCT06722326
Title: The Effects of 8-week Hydrogen-rich Water Consumption on Body Composition, Appetite and Obesity-specific Quality of Life, and Circulating Glucagon-like Peptide-1 in Obese Men and Women (Hydrappet): a Randomized Controlled Trial
Brief Title: Hydrogen-rich Water and Appetite in Obesity
Acronym: HYDRAPPET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Novi Sad, Faculty of Sport and Physical Education (Other)
Responsible Party: Principal Investigator, Sergej Ostojic, Professor and Head of the Lab, University of Novi Sad, Faculty of Sport and Physical Education
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 03-HRW-24
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: dihydrogen; appetite; LDL cholesterol; supplementation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen-rich water (Experimental): One liter per day of hydrogen rich water
  Interventions: Dietary Supplement: Dietary Supplement: Hydrogen-rich water
- Control water (Placebo Comparator): One liter per day of tap water
  Interventions: Dietary Supplement: Dietary Supplement: Control water

INTERVENTIONS:
Dietary Supplement: Dietary Supplement: Hydrogen-rich water — Hydrogen-rich water with 12 mg of hydrogen per serving
  Arms: Hydrogen-rich water
Dietary Supplement: Dietary Supplement: Control water — Control water with 0 mg of hydrogen per serving
  Arms: Control water

SUMMARY:
The main goal of this study is to investigate how dihydrogen supplementation impacts body composition, appetite, quality of life specific to obesity, and levels of the hormone GLP-1 in men and women with obesity. This randomized controlled trial aims to explore whether dihydrogen can improve these health indicators.

DETAILED DESCRIPTION:
The primary aim of this randomized controlled trial is to evaluate the effects of dihydrogen supplementation on body composition indices, appetite, obesity-specific quality of life, and circulating GLP-1 levels in obese men and women

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Body fat > 30% in women and > 25% in men
* Not physically active
* Informed consent signed

Exclusion Criteria:

* Major chronic disease and acute injuries
* History of dietary supplement use during the past 4 weeks
* History of obesity pharmaceuticals use during the past 8 weeks
* No consent to randomization
* Participation in other studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Appetite | Change from baseline appetite at 8 weeks
  Total scores for appetite as assessed by the the Food Cravings Questionnaire (FCQ)

SECONDARY OUTCOMES:
Obesity-related quality or life | Change from baseline total scores for obesity-related quality of life at 8 weeks
  Total scores for obesity-related quality of life as assessed by the The Impact of Weight on Quality of Life-Lite (IWQOL-Lite) questionnaire
Body fat | Change from baseline body fat at 8 weeks
  Percentage of body fat as assessed by a multifrequency bioelectrical impedance analyzer
Serum GLP-1 | Change from baseline GLP-1 at 8 weeks
  Serum levels of glucagon-like peptide-1 (GLP-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Bioenergetics Lab, Novi Sad, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in obesity. Data will be coded, with no PHI included. Approval of the request and execution of all applicable agreements are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Data obtained through this study may be provided to qualified researchers with academic interest in obesity.

REFERENCES:
- [Background] Korovljev D, Ostojic J, Todorovic N, Ostojic SM. Molecular hydrogen modulates brain glutamate/GABA-glutamine cycle in overweight humans. Arch Med Sci. 2023 Jul 13;19(4):1151-1153. doi: 10.5114/aoms/162938. eCollection 2023. PMID 37560746
- [Derived] Todorovic N, Baltic S, Nedeljkovic D, Kuzmanovic J, Korovljev D, Javorac D, Bijelic K, Kladar N, Tarnava A, Ostojic SM. The Effects of 8-Week Hydrogen-Rich Water Consumption on Appetite, Body Composition, Sleep Quality, and Circulating Glucagon-like Peptide-1 in Obese Men and Women (HYDRAPPET): A Randomized Controlled Trial. Medicina (Kaunas). 2025 Jul 18;61(7):1299. doi: 10.3390/medicina61071299. PMID 40731927